CLINICAL TRIAL: NCT06248151
Title: Acute Cardiovascular Responses to a Single Exercise Session in Patients With Post-Covid-19 Syndrome
Acronym: ExPostCovid-19
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Raphael Mendes Ritti Dias, Full Professor, University of Nove de Julho
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Acute_Covid; 0057/2022 (Other: CAPES)
Record Dates: First submitted 2024-02-06; First posted 2024-02-08 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Post-Acute COVID-19 Syndrome
Keywords: Post-Covid 19 Syndrome; Covid-19; fatigue; cardiovascular system; respiratory system; rehabilitation
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; COVID-19; Fatigue | interventions — Rehabilitation; Pliability

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): In the exercise session, participants will perform aerobic, free active and flexibility exercises and will last approximately 45 minutes.
  Interventions: Behavioral: Exercise session; Behavioral: Control session
- Control (Other): In the control session, participants will remain seated for 60 minutes.
  Interventions: Behavioral: Exercise session; Behavioral: Control session

INTERVENTIONS:
Behavioral: Exercise session — Session will included aerobic, resistance and flexibility exercises and will last approximately 45 minutes. The session will begin with aerobic exercises (5 min jumping jacks and 5 min stationary walking). Then, nine strength exercises will be performed for the main muscle groups (3 times of 12 to 15 repetitions, with a 1-minute rest interval) and finally stretching for the main muscle groups
  Other Names: Rehabilitation; Cardiorespiratory exercises; Resistance exercises; Flexibility
Behavioral: Control session — Remain seated for 60 min

SUMMARY:
The objective of the study is to compare the acute cardiorespiratory and perceptual responses to a physical exercise session in those infected by Covid-19 with and without persistent symptoms.

DETAILED DESCRIPTION:
The study will be a crossover carried out in two groups (with and without persistent symptoms of Covid-19). Participants in both groups will undergo a control session and an exercise session and cardiorespiratory and perceptual responses will be obtained before, during and after the sessions. In the exercise session, participants will perform aerobic exercises, strength exercises and muscle stretching, while in the control session participants will remain seated. Blood pressure, heart rate, cardiac autonomic modulation, peripheral oxygen saturation, vascular function and perception of affect will be obtained.

ELIGIBILITY:
Inclusion Criteria:

Post-Covid Syndrome group:

* have had a positive RT-PCR test for Covid-19;
* present persistent symptoms of Post Covid 19 syndrome, which have no other health explanation according to the criteria of the World Health Organization (WHO);
* have the cognitive and physical capacity to perform the exercises; It is
* low cardiovascular risk classification according to the American College of Sports Medicine criteria.

Healthy group:

* not present persistent symptoms of Post Covid 19 syndrome, which have no other health explanation according to the criteria of the World Health Organization (WHO);
* have the cognitive and physical capacity to perform the exercises; It is
* low cardiovascular risk classification according to the American College of Sports Medicine criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Change in Blood pressure | Before and 30 and 50 minutes after the end of the exercise and control interventions
  Assessment of the systolic and diastolic blood pressure using an automatic device
Change in Heart rate variability | Before and 30 and 50 minutes after the end of the exercise and control interventions
  Assessment of the heart rate variability indicators using a heart rate monitor
Change in flow mediated dilation | Before and 30 minutes after the end of the exercise and control interventions
  Assessment of the flow mediated dilation using a doppler ultrasound
Change in peak exhalation flow | Before and 5 minutes after the end of the exercise and control interventions
  Assessment of the peak exhalation flow using a peak flow device
Change in oxygen saturation | Before, during and 5 minutes after the end of the exercise and control interventions
  Assessment of the peripheral oxygen saturation using a pulse oximeter

SECONDARY OUTCOMES:
Change in heart rate | Before and continuously during exercise and control interventions
  Assessment of heart rate using a heart rate monitor
Change in affective response | Before and every 5 minutes during exercise and control interventions
  Assessment of affective response using a felling scale

CONTACTS AND LOCATIONS:
Overall Officials: Raphael Dias, PhD, Study Chair — University of Nove de Julho
Locations (1):
- Universidade Nove de Julho, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
Plan to share the data after completion upon resonable request